CLINICAL TRIAL: NCT00636909
Title: Nonmyeloablative Allogeneic Stem Cell Transplant for the Treatment of Hematologic Disorders
Brief Title: Nonmyeloablative Allo SCT for the Treatment of Hematologic Disorders
Acronym: MINI HEME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, David McDermott, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001P002293; W-99-0234-FB
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: AML; ALL; CML Chronic Phase, Accelerated Phase, or Blast Crisis; CLL; MDS; RELAPSED NON-HODGKIN'S OR HODGKIN'S LYMPHOMA; APLASTIC ANEMIA; MULTIPLE MYELOMA; MYELOPROLIFERATIVE DISORDER (P Vera, CMML, ET)
Keywords: AML; ALL; CML; CLL; MDS; NHL; HODGKIN'S LYMPHOMA; APLASTIC ANEMIA; MULTIPLE MYELOMA; MYELOPROLIFERATIVE DISORDER; ALLOGENEIC; STEM CELL TRANSPLANT; HEMATOLOGIC DISORDERS; CYCLOPHOSPHAMIDE; FLUDARABINE; CYCLOSPORINE; METHOTREXATE; G-CSF; GVHD; ENGRAFTMENT; CHIMERISM
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Blast Crisis; Anemia, Aplastic; Multiple Myeloma; Myeloproliferative Disorders; Hodgkin Disease; Hematologic Diseases | interventions — Cyclophosphamide; fludarabine; Cyclosporine; Methotrexate; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Study treatment arm with G-CSF
  Interventions: Drug: Cyclophosphamide; Drug: fludarabine; Drug: cyclosporine; Drug: methotrexate; Biological: G-CSF

INTERVENTIONS:
Drug: Cyclophosphamide — preparative cytoreduction
Drug: fludarabine — preparative cytoreduction
Drug: cyclosporine — immunosuppressive therapy
Drug: methotrexate — immunosuppressive therapy
Biological: G-CSF — foster engraftment

SUMMARY:
The purpose of this study is to provide allogeneic stem cell transplantation to patients who have not traditionally undergone this procedure because of it high incidence of treatment related side effects. We hope to decrease these side effects by decreasing the chemotherapy dose prior to transplant (non-myeloablative, smaller dose of chemotherapy given so bone marrow is not completely eliminated) and by using donated stem cells to treat cancer of the blood.

ELIGIBILITY:
Inclusion Criteria - Patient:

* AML, ALL,CML Chronic Phase, Accelerated Phase, or Blast Crisis, CLL, MDS, RELAPSED NON-HODGKIN'S OR HODGKIN'S LYMPHOMA, Aplastic Anemia, Multiple Myeloma, MYELOPROLIFERATIVE DISORDER (P Vera, CMML, ET
* Age less than 65 years
* Patients must have a healthy family member who is HLA-identical to the recipient or has 1 antigen mismatch and who is willing to receive a course of G-CSF and undergo 2-4 daily leukaphereses
* Each patient must sign an informed consent and be willing to participate as a research subject after having been advised of the nature and risk of the study prior to entering protocol

Inclusion Criteria - Donor:

* Absence of hematologic or marrow function related diseases that interferes with the collection of sufficient numbers of normal progenitor cells
* Absence of any medical condition that would pose a serious health risk by undergoing peripheral blood stem cell harvest
* Negative HIV, HTLV-1, Hepatitis B surface antigen and Hepatitis C
* The donor must be blood relation. A prospective related donor must be at least genotypically HLA-A, B, DR identical to the patient, but can differ for 1 HLA-locus.

Exclusion Criteria - Patient:

* Active CNS involvement
* Females who are pregnant or breast feeding
* ECOG performance status > 1. Karnofsky performance status < 80%
* LVEF < 40%
* Active viral, bacterial, or fungal infection
* Patients seropositive for HIV; HTLV -1
* Patients not providing informed consent
* Patients with known hypersensitivity to E. Coli derived product

Exclusion Criteria - Donor:

* A positive HIv infection or HTLV - 1 test or evidence of active/persistent viral hepatitis infection. Presence of any medical condition that would pose a serious health risk by undergoing peripheral blood stem cell harvest. Donors with known hypersensitivity to E. Coli derived products.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-07; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
durable engraftment | 100 days
hematopoeitic reconstitution | 3 years
evaluate the patterns of post-transplant chimerism among lymphoid and antigen presenting cells | 3 years

SECONDARY OUTCOMES:
disease free survival and overall survival | 3 years
incidence of treatment related toxicity and acute and chronic graft versus host disease | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: David F McDermott, MD, Principal Investigator — Beth Israel Deaconess Medical Center; David E Avigan, MD, Study Director — Beth Israel Deaconess Medical Center